CLINICAL TRIAL: NCT01230996
Title: A Phase I/II, Multi-Center Dose Escalation Study of Simultaneous Boost Intensity-Modulated Radiotherapy for Locally Advanced Cervical Cancer
Brief Title: Dose Escalation Study of Simultaneous Boost Intensity-Modulated Radiotherapy for Locally Advanced Cervical Cancer
Acronym: DEPICT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6867; ISRCTN76100993; NCT01793701 (obsolete NCT alias)
Record Dates: First submitted 2010-10-28; First posted 2010-10-29 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Locally Advanced Cervical Cancer
Keywords: cervical adenocarcinoma; cervical adenosquamous cell carcinoma; cervical squamous cell carcinoma; stage IB cervical cancer; stage IIA cervical cancer; stage IIB cervical cancer; stage III cervical cancer; stage IVA cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Radiotherapy, Intensity-Modulated; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose escalation study (Experimental): This is a dose escalation study of IMRT for women with locally advanced cervical cancer. Three dose levels will be investigated, (although, the first dose level is considered to be the equivalent to a standard pelvic dose with parametrial boost). Before moving to the next dose level it must be confirmed by the Chief Investigator that the Maximum Administrable Dose (MAD) has not been met in the previous dose level (see section 6.3). If MAD is reached before dose level 3 the study will stop. All patients enrolled on the study will undergo the same procedures at the same time points, regardless of the dose level they are being given (see section 5).
  Interventions: Drug: Cisplatin; Radiation: Intensity-modulated radiation therapy; Procedure: Intracavitary brachytherapy

INTERVENTIONS:
Drug: Cisplatin — Each patient will also receive chemotherapy with a drug called cisplatin, which is given intravenously through a drip in the arm once a week during their 6 week radiotherapy treatment. Again this is standard treatment for any patient with cervix cancer.
Radiation: Intensity-modulated radiation therapy — Patients in this trial will receive radiotherapy to the pelvic area with additional chemotherapy (chemoradiotherapy). This is the standard treatment for cervix cancer and will be almost identical to patients not taking part in this study. As patients in the study will be treated with IMRT, the total radiation dose will be slightly higher but without increasing the dose to normal tissue in the pelvis. This will mean the number of radiotherapy treatments that each patient receives in the study is between 27 and 30 compared with the usual 28. Each patient will undergo 6 weeks of radiotherapy treatment and must attend the radiotherapy department hospital once daily (Monday to Friday) over 6 weeks. Each treatment lasts for approximately 10 15 minutes. This is exactly the same as standard practice if patients were not participating in the trial.
  Other Names: IMRT
Procedure: Intracavitary brachytherapy — Intracavitary brachytherapy Intracavitary brachytherapy will be given towards the end of external beam radiotherapy usually weeks five and six. This is routine treatment and will be given according to local practice As is the convention patients will be reviewed weekly (more frequently if necessary) by their study doctor and will have weekly blood tests to measure full blood count and urea and electrolytes.

SUMMARY:
This will be the first study to assess the clinical feasibility of dose escalation with simultaneous integrated boost intensity-modulated radiotherapy for patients with locally advanced cervical cancer. Following screening to confirm eligibility patients will commence a six week treatment period. After this, patients will be followed up by visits to clinic every 3 months for a period of 24 months (2 years). End of study is defined as 24 months after treatment. Patients will be followed up for a minimum of 5 years (as per local policy) after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed squamous cell carcinoma, adenocarcinoma or poorly differentiated carcinoma of the cervix
2. FIGO stage IIB-IVA (any pelvic nodal status) and FIGO stage 1B2 and IIA with pelvic nodal involvement
3. Measurable disease on MRI
4. Age > 18 years (no upper limit)
5. WHO performance status 0,1
6. Adequate renal function with EDTA clearance> 55ml/min
7. Adequate liver function, as defined by ALT or AST less than 2.5 x ULN, and bilirubin less than 1.25 x ULN
8. Adequate bone marrow function, defined by WCC >3.0 x 109/litre, neutrophils > 1.5 x 109/litre and platelets > 100 x 109 /litre
9. Able to understand and give written informed consent

Exclusion Criteria:

1. Evidence of common iliac or para-aortic nodal involvement, or distant metastases
2. Previous history of cancer except skin tumour
3. Previous pelvic radiotherapy or surgery other than toparoscopic node disection
4. Previous history of pelvic adhesions, inflammatory bowel disease, pelvic inflammatory disease or diabetes mellitus
5. Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for protocol therapy if required. Acceptable contraception should be used such as barrier or hormonal methods.
6. Females must not be pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Grade 3 gastrointestinal toxicity at 6 months as defined by CTCAE v 3.0 | 6 months

SECONDARY OUTCOMES:
Response rate assessed radiologically at 3 and 12 months | 3 and 12 months
Local control of the disease at 2 years | 2 years
Late toxicity at 2 years as defined by CTCAE v 3.0 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Powell, Principal Investigator — Barts & The London NHS Trust
Locations (4):
- United Kingdom (4):
  - Saint Bartholomew's Hospital, London, England
  - Hammersmith Hospital, London, England
  - Royal Marsden - London, London, England
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield